CLINICAL TRIAL: NCT07306767
Title: Role of Ultrasound Estimation of Intra-Vesical Prostatic Protrusion in Predicting the Response to Medical Therapy in Patients With Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia
Brief Title: Ultrasound IPP to Predict Response to Medical Therapy in LUTS/BPH
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mustafa mohamed esmail aboalmagd, Resident of Urology, Ain Shams University
Other Study IDs: FMASU_MS403_2025
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms; Bladder Outlet Obstruction
Keywords: Intravesical prostatic protrusion; Transabdominal ultrasound; Prostate ultrasound; International Prostate Symptom Score; Quality of life; Uroflowmetry; Maximum urinary flow rate; Post-void residual urine; Detrusor wall thickness
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms; Urinary Bladder Neck Obstruction | interventions — Adrenergic alpha-Antagonists; 5-alpha Reductase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- IPP Grade I (<5 mm): Participants with lower urinary tract symptoms secondary to benign prostatic hyperplasia and intravesical prostatic protrusion less than 5 millimetres measured by transabdominal ultrasonography at bladder volume 100-200 millilitres. Participants received medical therapy as prescribed by the treating urologist and were followed for 6 months with assessments at baseline, 3 months, and 6 months including International Prostate Symptom Score/quality of life, uroflowmetry, and ultrasound parameters.
  Interventions: Diagnostic Test: Transabdominal ultrasound measurement of intravesical prostatic protrusion; Drug: Alpha-adrenergic blocker; Drug: 5-alpha reductase inhibitor
- IPP Grade II (5-10 mm): Participants with lower urinary tract symptoms secondary to benign prostatic hyperplasia and intravesical prostatic protrusion 5 to 10 millimetres measured by transabdominal ultrasonography at bladder volume 100-200 millilitres. Participants received medical therapy as prescribed by the treating urologist and were followed for 6 months with assessments at baseline, 3 months, and 6 months including International Prostate Symptom Score/quality of life, uroflowmetry, and ultrasound parameters.
  Interventions: Diagnostic Test: Transabdominal ultrasound measurement of intravesical prostatic protrusion; Drug: Alpha-adrenergic blocker; Drug: 5-alpha reductase inhibitor
- IPP Grade III (>10 mm): Participants with lower urinary tract symptoms secondary to benign prostatic hyperplasia and intravesical prostatic protrusion greater than 10 millimetres measured by transabdominal ultrasonography at bladder volume 100-200 millilitres. Participants received medical therapy as prescribed by the treating urologist and were followed for 6 months with assessments at baseline, 3 months, and 6 months including International Prostate Symptom Score/quality of life, uroflowmetry, and ultrasound parameters.
  Interventions: Diagnostic Test: Transabdominal ultrasound measurement of intravesical prostatic protrusion; Drug: Alpha-adrenergic blocker; Drug: 5-alpha reductase inhibitor

INTERVENTIONS:
Diagnostic Test: Transabdominal ultrasound measurement of intravesical prostatic protrusion — Transabdominal ultrasonography; TAUS; Ultrasound IPP measurement Intervention Description: Intravesical prostatic protrusion was measured using transabdominal ultrasonography in the midsagittal plane at a bladder volume of approximately 100-200 millilitres. The measurement was defined as the distance (millimetres) from the bladder neck to the tip of the protruding prostatic tissue, and participants were categorized into Grade I (<5 millimetres), Grade II (5-10 millimetres), or Grade III (>10 millimetres). Ultrasound assessment was performed at baseline and during follow-up per protocol.
Drug: Alpha-adrenergic blocker — Participants received an alpha-adrenergic blocker as part of standard medical therapy for benign prostatic hyperplasia-related lower urinary tract symptoms. The specific agent, dose, dosing frequency, and duration were prescribed by the treating urologist and recorded throughout follow-up.
Drug: 5-alpha reductase inhibitor — Participants received a 5-alpha reductase inhibitor as part of standard medical therapy for benign prostatic hyperplasia-related lower urinary tract symptoms. The specific agent, dose, dosing frequency, and duration were prescribed by the treating urologist and recorded throughout follow-up.

SUMMARY:
This prospective cohort study evaluated whether transabdominal ultrasound measurement of intravesical prostatic protrusion predicts symptom severity and response to medical therapy in men aged 50 years or older with lower urinary tract symptoms secondary to benign prostatic hyperplasia. At baseline, participants underwent clinical evaluation, laboratory assessment including prostate-specific antigen, symptom scoring using the International Prostate Symptom Score and quality of life index, uroflowmetry, and transabdominal ultrasonography to measure prostate volume, bladder parameters, post-void residual urine, detrusor wall thickness, and intravesical prostatic protrusion. Participants were grouped by intravesical prostatic protrusion grade (less than 5 millimetres, 5 to 10 millimetres, and greater than 10 millimetres) and were followed for six months with reassessments at three and six months to evaluate response to medical therapy and identify patients who required escalation of treatment or surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male participants aged 50 years or older.
* Lower urinary tract symptoms secondary to benign prostatic hyperplasia.
* Moderate to severe symptoms with International Prostate Symptom Score 15 to 35.
* Prostate volume 30 to 100 millilitres.
* Maximum urinary flow rate less than 15 millilitres per second.
* No hydronephrosis due to bladder outlet obstruction.
* Normal prostate-specific antigen or normal free-to-total prostate-specific antigen ratio.

Exclusion Criteria:

* History of prostate, bladder, or lower urinary tract surgery.
* Neurological disease affecting lower urinary tract function.
* Active urinary tract infection and/or symptomatic urinary tract stones.
* Post-void residual urine volume greater than 200 millilitres.
* Urethral stricture.
* Prostate cancer or bladder cancer.

Min Age: 50 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Men aged 50 years or older with moderate to severe lower urinary tract symptoms secondary to benign prostatic hyperplasia attending urology outpatient services at Ain Shams University Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Change in International Prostate Symptom Score | Baseline and 6 months
  The International Prostate Symptom Score was used to quantify lower urinary tract symptom severity. The outcome was the change in total score between baseline (pre-treatment) and the 6-month follow-up visit.

SECONDARY OUTCOMES:
Change in quality of life score | Baseline and 6 months
  Change in the quality of life index associated with the International Prostate Symptom Score between baseline and 6 months.
Change in maximum urinary flow rate | Baseline and 6 months
  Change in maximum urinary flow rate measured by uroflowmetry between baseline and 6 months.
Change in post-void residual urine volume | Baseline and 6 months
  Change in post-void residual urine volume measured by transabdominal ultrasonography between baseline and 6 months.
Change in detrusor wall thickness | Baseline and 6 months
  Change in detrusor wall thickness measured by transabdominal ultrasonography between baseline and 6 months.
Need for escalation of management during follow-up | Up to 6 months
  Proportion of participants who required escalation of management during follow-up (for example, change or intensification of medical therapy or referral for surgical management) due to persistent symptoms or poor objective improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data collected during the study will be shared, including baseline and follow-up measurements (International Prostate Symptom Score and quality of life index, uroflowmetry parameters, transabdominal ultrasound parameters including intravesical prostatic protrusion, prostate volume, post-void residual urine, and detrusor wall thickness), along with a data dictionary. Direct identifiers will be removed and data will be coded prior to sharing.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: De-identified data will be available beginning 6 months after study completion and will remain available for 5 years.
Access Criteria: Data will be shared with qualified researchers upon reasonable request and after review and approval by the study investigators and the institutional administration. Requesters must submit a proposal outlining objectives and planned analyses and must sign a data use agreement that prohibits re-identification and limits use to the approved purpose.